CLINICAL TRIAL: NCT05242341
Title: A Randomized Controlled Trial to Explore Whether the Patients With Cancers on Clinical Trials Can Use the Health Insurance APP-My Health Bank to Increase Understanding and Safety of Treatment
Brief Title: Increase Understanding and Safety of Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202106191RINA
Record Dates: First submitted 2021-08-08; First posted 2022-02-16 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Hematology; Oncology
Keywords: randomized controlled trial; application(APP); My health bank
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- app use teaching (Experimental): Intervention includes teach the subjects one-on-one to use the "My Health Bank" for 30 minutes (such as download, register, test, find information, etc.), and provide pre-recorded 1-minute instructional videos for viewing when needed at home. The intervention group also accepts to follow the use of My Health Bank app at home every two weeks for a period of two months. Both groups will receive pre- and post-evaluations, including knowledge of the disease, understanding of lab data, and knowledge of medication safety (prohibited medicines and concomitant medications).
  Interventions: Behavioral: application(APP) teaching
- B (No Intervention): will receive pre- and post-evaluations, including knowledge of the disease, understanding of lab data, and knowledge of medication safety

INTERVENTIONS:
Behavioral: application(APP) teaching — Teaching the use of the APP
  Arms: app use teaching

SUMMARY:
Purpose: The purpose of this study is to use a randomized controlled trial to explore whether the patients with cancers on clinical trials can use the Health Insurance APP-My Health Bank to increase understanding and safety of treatment. It is of hope that the results of this study can help confirm whether cancer patients participate in clinical trials, learn to use the " Health Insurance APP-My Health Bank ", can increase the safety of treatment, including the understanding of the disease , the understanding of the lab data, and the communication about contraindications and concurrent use of medications. The results of this research will help clinical healthcare professionals promote the use of My Health Bank, and improve the safety of clinical trials, as well as to increase the communications between patients, doctors and nurses.

Methods: In this study, cancer patients (hematology-oncology patients are the priority invitations) were invited to participate in clinical trials in the outpatient and inpatient units. After explaining that they agreed to participate in the study, they were randomlyassigned to the experimental group and the control group. Intervention includes teach the subjects one-on-one to use the "My Health Bank" for 30 minutes (such as download, register, test, find information, etc.), and provide pre-recorded 1-minute instructional videos for viewing when needed at home. The intervention group also accepts to follow the use of My Health Bank app at home every two weeks for a period of two months. Both groups will receive pre- and post-evaluations, including knowledge of the disease, understanding of lab data, and knowledge of medication safety (prohibited medicines and concomitant medications). Post-intervention, the intervention group will also be evaluated on the "Satisfaction and Quality of Technology Use" of My Health Bank APP. Data analysis is expected to adopt Intention-to-treat analysis (ITT) method to compare the differences before and after intervention between the two groups to verify teach patients the clinical feasibility of using a My Health Bank and the effect of assisting patient care.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 20, the subject voluntarily accepts this study and signs the consent form
* Participants in clinical trials of hematological tumor-related diseases (have been or are participating in it)
* Need to be literate and can communicate in Chinese and Taiwanese
* Have a mobile phone or electronic device to download the my health bank APP and be willing to cooperate with it for at least two months of continuous use

Exclusion Criteria:

* I have downloaded the "my health bank APP" and use well
* Cognitive impairment diseases (e.g. dementia)
* The clinical trial protocol that originally participated in that it is not allowed to articipate in other interventional studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Drug safety and knowledge of diseases and app satisfaction | 2 months
  The Questionnaire include two scale, the first one is the scale of drug safety and knowledge of diseases , the minimum score is 8 points and the maximum is 40 points, higher scores mean a better outcome; the second scale is for app satisfaction, the minimum score is 0 point and the maximum is 55 points, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Chen Chang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided